CLINICAL TRIAL: NCT04185831
Title: MEGALiT - a Multicenter, Basket and Umbrella Explorative Trial on the Efficacy and Safety of Molecular Profile Selected Commercially Available Targeted Anti-cancer Drugs in Patients With Advanced Cancers Progressive on Standard Therapy
Brief Title: A MolEcularly Guided Anti-Cancer Drug Off-Label Trial
Acronym: MEGALiT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Nygren, MD, PhD, professor in oncology, Uppsala University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEGALiT1901
Record Dates: First submitted 2019-11-08; First posted 2019-12-04 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor
Keywords: mutation status; mutational burden; molecular profiling; precision medicine
MeSH Terms: interventions — atezolizumab; Everolimus; cobimetinib; niraparib

STUDY DESIGN:
Intervention Model Description: Combined umbrella and basket trial. Treatment selection based on mutation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NF1/MAP2K1 (Experimental): Cobimetinib, 60mg po daily. 28 day cycle; day 1-21 60mg daily, day 22-28 rest period.
  Interventions: Drug: Cobimetinib
- MTOR/TSC1/TSC2 (Experimental): Everolimus, 10mg po daily.
  Interventions: Drug: Everolimus
- Mutation burden (Experimental): Atezolizumab. 1200mg iv every 3 weeks.
  Interventions: Drug: Atezolizumab
- PPARi (Experimental): Niraparib. 300mg po daily.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Atezolizumab — PD-L1 inhibitor
  Other Names: Tecentriq
  Arms: Mutation burden
Drug: Everolimus — MTOR inhibitor
  Other Names: Afinitor
  Arms: MTOR/TSC1/TSC2
Drug: Cobimetinib — MEK inhibitor
  Other Names: Cotellic
  Arms: NF1/MAP2K1
Drug: Niraparib — PARP inhibitor
  Other Names: Zejula
  Arms: PPARi

SUMMARY:
This is a prospective, open-label, non-randomized combined basket- and umbrella trial divided in two parts; a limited feasibility-oriented part 1 including 154 patients and 3 treatment cohorts and part 2 that will include an expanded cohort of patients and treatment cohorts. The overall aims of the study are to test the feasibility, safety and efficacy of comprehensive genomic profiling on fresh tumor biopsies as a basis for treatment decision making and to compare two different sequencing, bioinformatics and decision-making platforms (part 1). Also to evaluate the efficacy and safety of off-label treatment with cancer drugs in patients selected based on genomic biomarker matching.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized combined basket- and umbrella trial divided in two parts; a limited feasibility-oriented part 1 including 154 patients and 3 treatment cohorts (mutation/drug) and part 2 that will include an expanded cohort of patients and treatment cohorts. The overall aims of the study are to test the feasibility, safety and efficacy of comprehensive genomic profiling on fresh tumor biopsies as a basis for treatment decision making and to compare two different sequencing, bioinformatics and decision-making platforms (part 1). Also to evaluate the efficacy and safety of off-label treatment with cancer drugs in patients selected based on genomic biomarker matching.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age >18 years)
2. Patients with histologically-proven, locally advanced or metastatic solid tumor (part 1; hematological malignancies also eligible in part 2) progressive while on last line established therapy considered available for the patient. For re-recruitment (part 2) patients must be progressive while on trial defined treatment or off-protocol treatment.
3. Fresh tumor sampling by biopsy must be possible, except for patients with CNS malignancy who can be included based on molecular analysis of archived tumor material.
4. ECOG performance status 0-2.
5. Patients must have acceptable organ function as defined below:

   1. Absolute neutrophil count ≥ 1.5 x 10^9/L
   2. Hemoglobin > 90 g/L
   3. Platelets > 75 x 10^9/L
   4. Total bilirubin < 2 x ULN
   5. ASAT (SGOT) and ALAT (SGPT) < 2.5 x institutional ULN (or < 5 x ULN in patients with known hepatic metastases)
   6. Serum creatinine ≤ 1.5 × ULN or calculated or measured creatinine clearance ≥ 50 mL/min/1.73 m2
6. Patients must have objectively measurable disease (by physical or radiographic examination).
7. Ability to understand and the willingness to sign a written informed consent document.
8. For orally administered drugs, the patient must be able to swallow and tolerate oral medication and must have no known malabsorption syndrome.
9. Negative pregnancy test in women of childbearing potential (premenopausal or <12 months of amenorrhea post-menopause and who have not undergone surgical sterilization). Women of childbearing potential must use highly effective method of contraception, i.e. combined hormonal contraception, or progestogen-only hormonal contraception, or intrauterine device, or intrauterine hormone-releasing system, or bilateral tubal occlusion, or vasectomized partner, or sexual abstinence for the duration of participation in the study, and four months following completion of study therapy.
10. Selected tumor types might have disease-specific inclusion criteria, defined by disease-specific study appendix.

Exclusion Criteria:

1. Ongoing treatment-related toxicity > grade 2.
2. Patients receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g., megestrol acetate, bisphosphonates, somatostatin analogues and prednisone, or equivalent, >5 mg/d). These medications must have been started ≥ 1 week prior to the screening visit on this study. Radiotherapy to non-target lesions is allowed.
3. Patients pregnant or nursing.
4. Patients of childbearing potential and sexually active and not willing to use highly effective contraceptive.
5. Patients with known active progressive CNS metastases. Patients with previously treated CNS metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within the 3 months prior to inclusion. All patients with previously treated CNS metastases must be stable for at least 1 month after completion of treatment and off steroid treatment prior to inclusion.
6. Some concomitant diseases qualified for exclusion as detailed in main protocol.
7. Other serious underlying medical conditions, which, in the Investigator's judgment, could impair the ability of the patient to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) and tumor control rate [Time Frame: From first dose up to 24 months] | 1 year follow-up after LPFV
  The proportion of patients that have a best overall response of complete response (CR), partial response (PR) or stable disease ≥16 weeks, as assessed by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Additional measurements of treatment efficacy | 1 year follow-up after LPFV
  Time to and duration of tumor response and stable disease, progression free survival, overall survival and progression free survival on study drug compared with that on the treatment preceding study drug treatment.
Drug-related safety, evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03 | 1 year follow-up after LPFV
  Incidence and severity of study drug related adverse events (AEs) and serious adverse events (SAEs). Include recording of changes in laboratory values, vital signs (body temperature, blood pressure, heart rate, respiratory rate), and assessment of physical, dermatological examinations graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
Biopsy safety: NCI Common Terminology Criteria for Adverse Events 4.03 as grade 3 - 4 adverse event related to the procedure | 1 year follow-up after LPFV
  Safety of core needle biopsy in advanced cancer scored according to NCI Common Terminology Criteria for Adverse Events 4.03 as grade 3 - 4 adverse event related to the procedure.
Genomic analysis | 1 year follow-up after LPFV
  Actionable target concordance between genomic analysis results from the Foundation Medicine platform F1CDx with that from the similar local analysis.
Overall survival | 1 year follow-up after LPFV
  Overall survival of patients starting treatment in accordance with 1 of the 4 groups of genomic markers compared with patients included in the trial but that do not start such treatment due to lack of appropriate marker.
Feasibility of study design | 1 year follow-up after LPFV
  Feasibility of comprehensive genomic testing of fresh tumor tissue for treatment decision, defined as the proportion of patients included with actionable genomic analysis within 4 weeks from inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nygren, MD, PhD, Principal Investigator — Uppsala University Hospital; Peter Asplund, BSc, Study Director — Uppsala University Hospital
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Uppsala University Hospital, Uppsala